CLINICAL TRIAL: NCT03113136
Title: Examination of Low Wattage and High Wattage E-Cigarettes
Acronym: SWITCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH); University of Minnesota (Other)
Responsible Party: Principal Investigator, Theodore Wagener, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: OSU-19095; R01CA204891-01 (NIH); NCI-2019-01855 (Registry Identifier: CTRP (Clinical Trial Reporting Program)
Record Dates: First submitted 2017-03-22; First posted 2017-04-13 (Actual); Results first posted 2024-02-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Smoking, Cigarette; Smoking, Tobacco; Nicotine Dependence; Exposure to Toxic Agent
MeSH Terms: conditions — Cigarette Smoking; Tobacco Smoking; Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low wattage E cigarette device (Active Comparator)
  Interventions: Behavioral: Low wattage E cigarette device
- High wattage E cigarette device (Active Comparator)
  Interventions: Behavioral: High wattage E cigarette device
- Usual brand cigarette (Active Comparator)
  Interventions: Behavioral: Usual brand cigarette

INTERVENTIONS:
Behavioral: Low wattage E cigarette device — The low wattage E cigarette device will be provided to the participant and they will be instructed to vape ad libitum for 12 weeks and then be assessed at 6 months and 12 months for continued use of device.
  Arms: Low wattage E cigarette device
Behavioral: High wattage E cigarette device — The high wattage E cigarette device will be provided to the participant and they will be instructed to vape ad libitum for 12 weeks and then be assessed at 6 months and 12 months for continued use of device.
  Arms: High wattage E cigarette device
Behavioral: Usual brand cigarette — The usual brand of cigarettes will be provided to the participant and they will be instructed to smoke ad libitum for the duration of the study.
  Arms: Usual brand cigarette

SUMMARY:
The overall aim of the proposed study is to evaluate the effect of switching from conventional cigarettes to either a LWe or HWe on smoking behavior, product use patterns and continued use, as well as biomarkers of toxicant exposure and effects.

ELIGIBILITY:
Inclusion Criteria:

1. smoke ≥5 cigarettes per day for the past year;
2. no quit attempt in the prior 3 months and no plan to quit in the next 3 months;
3. read, write, and speak in English;
4. report at least minimal interest in switching to an alternative product (> "not at all" on a Likert scale);
5. never purchased or regularly used a tank system, mechanical mod, or advanced personal vaporizer EC, though previous use of cig-a-like devices will be allowed but not in the last 3 months;
6. plan to live in the local area for next year; and
7. have reliable means of transport. -

Exclusion Criteria:

1. <18 years old;
2. unstable or significant medical condition such as respiratory, kidney, or liver disease that could potentially affect biomarker data;
3. unstable or significant psychiatric conditions (past and stable conditions will be allowed);
4. history of cardiac event or distress within the past 3 months; and
5. currently pregnant, planning to become pregnant, or breastfeeding (n.b: pregnancy status will continue to be evaluated throughout the study at each visit).

   -

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Wagener, PhD, Principal Investigator — Ohio State Comprehensive Cancer Center
Locations (1):
- The Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Brand Cigarette | Low Wattage E Cigarette Device | High Wattage E Cigarette Device
Started | 105 | 133 | 134
Week 1 | 101 | 115 | 122
Week 4 | 99 | 97 | 113
Week 8 | 98 | 86 | 94
Week 12 | 95 | 84 | 92
Week 26 | 77 | 69 | 73
Week 52 | 78 | 67 | 65
Completed | 78 | 67 | 65
Not Completed | 27 | 66 | 69
Not completed — Lost to Follow-up | 22 | 47 | 54
Not completed — Withdrawal by Subject | 4 | 13 | 14
Not completed — Ineligible | 0 | 2 | 1
Not completed — Study Team Decision | 1 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Brand Cigarette | Low Wattage E Cigarette Device | High Wattage E Cigarette Device | Total
Number analyzed (Participants) | 105 | 133 | 134 | 372
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.95 (10.99) | 39.69 (11.05) | 40.47 (11.13) | 40.33 (11.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 81 | 84 | 233
  Male | 37 | 52 | 50 | 139
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 2 | 5
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 13 | 13 | 10 | 36
  White | 80 | 101 | 113 | 294
  More than one race | 6 | 13 | 7 | 26
  Unknown or Not Reported | 3 | 4 | 2 | 9
Cigarettes Smoked per Day [Mean (Standard Deviation); unit: cigarettes per day] — Population: 3 participants were missing data on the number of cigarettes smoked per day at baseline.
  cigarettes per day
    number analyzed (Participants) | 103 | 133 | 133 | 369
    (all) | 18.13 (9.11) | 16.86 (9.10) | 17.33 (8.65) | 17.38 (8.93)

OUTCOME MEASURES:

1. Primary Outcome: Complete Change From Conventional Cigarettes - Self Report
Description: Self-Reported 7-day Point Prevalence Abstinence from Cigarettes evaluated via the Timeline Follow Back Questionnaire.
  An intent-to-treat approach is taken where no participants are excluded and missing data is imputed as not abstinent from cigarettes.
Time Frame: Week 4, Week 8, Week 12, Week 26, and Week 52
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Brand Cigarette | Low Wattage E Cigarette Device | High Wattage E Cigarette Device
Number analyzed (Participants) | 105 | 133 | 134
Participants
  Week 4 | 0 | 12 | 10
  Week 8 | 0 | 19 | 10
  Week 12 | 0 | 16 | 16
  Week 26 | 5 | 20 | 9
  Week 52 | 4 | 13 | 8

2. Primary Outcome: Complete Change From Conventional Cigarettes - Biochemically Verified
Description: Intent to treat biochemically verified abstinence rates - participants reporting both 7-day point prevalence abstinence and an exhaled carbon monoxide reading less than or equal to 10.
  An intent-to-treat approach is taken where no participants are excluded and missing data is imputed as not abstinent from cigarettes.
Time Frame: Week 4, Week 8, Week 12, Week 26, and Week 52
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Brand Cigarette | Low Wattage E Cigarette Device | High Wattage E Cigarette Device
Number analyzed (Participants) | 105 | 133 | 134
Participants
  Week 4 | 0 | 10 | 9
  Week 8 | 0 | 16 | 8
  Week 12 | 0 | 15 | 11
  Week 26 | 5 | 18 | 6
  Week 52 | 4 | 11 | 8

3. Secondary Outcome: Cigarette Dependence
Description: Cigarette Dependence Scale Scores range from 12 to 60 with higher scores indicating greater dependence.
Time Frame: Baseline, Week 1, Week 4, Week 8, Week 12, Week 26 and Week 52
Population: Participants who attended the study visit and responded to the items in the cigarette dependence scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Brand Cigarette | Low Wattage E Cigarette Device | High Wattage E Cigarette Device
Number analyzed (Participants) | 105 | 133 | 134
score on a scale
  Baseline: number analyzed (Participants) | 98 | 125 | 127
  Baseline | 48.27 (7.36) | 47.63 (7.51) | 47.45 (8.79)
  Week 1: number analyzed (Participants) | 93 | 98 | 99
  Week 1 | 48.45 (6.96) | 43.71 (8.70) | 43.33 (9.05)
  Week 4: number analyzed (Participants) | 89 | 75 | 94
  Week 4 | 48.90 (7.57) | 41.89 (9.74) | 40.21 (10.13)
  Week 8: number analyzed (Participants) | 96 | 60 | 87
  Week 8 | 48.27 (8.06) | 41.80 (9.14) | 40.06 (10.68)
  Week 12: number analyzed (Participants) | 93 | 62 | 74
  Week 12 | 48.03 (7.78) | 41.32 (9.67) | 40.84 (9.59)
  Week 26: number analyzed (Participants) | 76 | 52 | 66
  Week 26 | 47.00 (8.72) | 40.67 (11.27) | 41.15 (9.57)
  Week 52: number analyzed (Participants) | 60 | 44 | 73
  Week 52 | 45.03 (9.74) | 42.32 (11.05) | 41.26 (10.36)

4. Secondary Outcome: Cigarette Likeability/Preference
Description: Cigarette Evaluation Scale Scores range from 1 to 7 with higher scores indicating greater satisfaction, psychological reward, aversion, or relief
Time Frame: Baseline, Week 4, Week 12, Week 26, and Week 52
Population: Participants who attended the study visit and answered the Cigarette Evaluation Scale items
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Brand Cigarette | Low Wattage E Cigarette Device | High Wattage E Cigarette Device
Number analyzed (Participants) | 105 | 133 | 134
score on a scale
  Satisfaction - Baseline | 4.68 (1.17) | 5.01 (1.27) | 4.81 (1.28)
  Psychological Reward - Baseline: number analyzed (Participants) | 104 | 133 | 134
  Psychological Reward - Baseline | 4.30 (1.13) | 4.54 (1.36) | 4.13 (1.49)
  Aversion - Baseline: number analyzed (Participants) | 105 | 132 | 133
  Aversion - Baseline | 2.44 (0.90) | 2.13 (0.80) | 2.16 (0.89)
  Relief - Baseline: number analyzed (Participants) | 105 | 132 | 133
  Relief - Baseline | 5.39 (0.94) | 5.19 (1.03) | 5.15 (0.93)
  Satisfaction - Week 4: number analyzed (Participants) | 99 | 116 | 122
  Satisfaction - Week 4 | 4.68 (1.38) | 4.63 (1.50) | 4.39 (1.40)
  Psychological Reward - Week 4: number analyzed (Participants) | 99 | 116 | 123
  Psychological Reward - Week 4 | 4.18 (1.19) | 4.09 (1.41) | 3.62 (1.50)
  Aversion - Week 4: number analyzed (Participants) | 99 | 116 | 122
  Aversion - Week 4 | 2.25 (0.90) | 2.28 (0.86) | 2.43 (0.91)
  Relief - Week 4: number analyzed (Participants) | 98 | 115 | 121
  Relief - Week 4 | 5.38 (0.97) | 5.19 (1.06) | 4.88 (1.10)
  Satisfaction - Week 12: number analyzed (Participants) | 98 | 96 | 108
  Satisfaction - Week 12 | 4.74 (1.50) | 4.26 (1.61) | 4.27 (1.68)
  Psychological Reward - Week 12: number analyzed (Participants) | 98 | 97 | 108
  Psychological Reward - Week 12 | 4.02 (1.38) | 3.72 (1.60) | 3.61 (1.49)
  Aversion - Week 12: number analyzed (Participants) | 97 | 98 | 107
  Aversion - Week 12 | 2.35 (1.01) | 2.40 (0.96) | 2.45 (0.95)
  Relief - Week 12: number analyzed (Participants) | 97 | 96 | 108
  Relief - Week 12 | 5.26 (1.04) | 5.26 (1.08) | 4.88 (1.14)
  Satisfaction - Week 26: number analyzed (Participants) | 84 | 83 | 98
  Satisfaction - Week 26 | 4.47 (1.51) | 4.23 (1.68) | 4.26 (1.57)
  Psychological Reward - Week 26: number analyzed (Participants) | 84 | 83 | 98
  Psychological Reward - Week 26 | 3.92 (1.38) | 3.69 (1.51) | 3.53 (1.42)
  Aversion - Week 26: number analyzed (Participants) | 83 | 83 | 98
  Aversion - Week 26 | 2.33 (0.94) | 2.46 (0.97) | 2.36 (0.92)
  Relief - Week 26: number analyzed (Participants) | 84 | 81 | 97
  Relief - Week 26 | 5.23 (1.08) | 5.22 (1.06) | 4.89 (1.09)
  Satisfaction - Week 52: number analyzed (Participants) | 64 | 62 | 94
  Satisfaction - Week 52 | 4.27 (1.50) | 4.17 (1.71) | 4.37 (1.55)
  Psychological Reward - Week 52: number analyzed (Participants) | 63 | 62 | 94
  Psychological Reward - Week 52 | 3.70 (1.41) | 3.74 (1.50) | 3.59 (1.57)
  Aversion - Week 52: number analyzed (Participants) | 64 | 62 | 94
  Aversion - Week 52 | 2.32 (1.00) | 2.68 (1.07) | 2.42 (0.89)
  Relief - Week 52: number analyzed (Participants) | 64 | 62 | 94
  Relief - Week 52 | 5.26 (1.23) | 4.96 (1.18) | 4.84 (1.16)

5. Secondary Outcome: EC Likeability/Preference
Description: EC modified-Cigarette Evaluation Scale Scores range from 1 to 7 with higher scores indicating greater satisfaction, psychological reward, aversion, or relief.
  No results are reported for the Usual Brand Cigarette arm as the participants in this arm did not receive a study e-cigarette device and thus were not asked to respond to the e-cigarette modified cigarette evaluation scale items.
Time Frame: Week 4, Week 12
Population: Participants who attended the study visit and answered the EC modified Cigarette Evaluation Scale items
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Wattage E Cigarette Device | High Wattage E Cigarette Device
Number analyzed (Participants) | 133 | 134
score on a scale
  Satisfaction - Week 4: number analyzed (Participants) | 109 | 115
  Satisfaction - Week 4 | 4.67 (1.28) | 4.63 (1.50)
  Psychological Reward - Week 4: number analyzed (Participants) | 109 | 117
  Psychological Reward - Week 4 | 2.93 (1.26) | 2.61 (1.33)
  Aversion - Week 4: number analyzed (Participants) | 109 | 117
  Aversion - Week 4 | 1.48 (0.60) | 1.50 (0.67)
  Relief - Week 4: number analyzed (Participants) | 108 | 117
  Relief - Week 4 | 4.21 (1.40) | 4.06 (1.33)
  Satisfaction - Week 12: number analyzed (Participants) | 92 | 103
  Satisfaction - Week 12 | 4.44 (1.47) | 4.65 (1.61)
  Psychological Reward - Week 12: number analyzed (Participants) | 92 | 102
  Psychological Reward - Week 12 | 2.73 (1.41) | 2.66 (1.37)
  Aversion - Week 12: number analyzed (Participants) | 92 | 103
  Aversion - Week 12 | 1.40 (0.55) | 1.46 (0.72)
  Relief - Week 12: number analyzed (Participants) | 93 | 103
  Relief - Week 12 | 4.18 (1.38) | 4.13 (1.41)

6. Secondary Outcome: EC Abuse Liability
Description: An adapted version of the Drug Effects/Liking Questionnaire will assess the desire and liking of all three study products. Five visual analog scale items ranging from 0 ('not at all') to 100 ('extremely') assessed wanting to smoke the product again, liking the product, enjoying the product, finding the product pleasurable and satisfying.
Time Frame: Week 4, Week 12, Week 26, and Week 52
Population: For weeks 26 and 52, only participants who reported continued use of the study product were asked the items on the questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Brand Cigarette | Low Wattage E Cigarette Device | High Wattage E Cigarette Device
Number analyzed (Participants) | 105 | 133 | 134
score on a scale
  Want - Week 4: number analyzed (Participants) | 100 | 110 | 114
  Want - Week 4 | 72.08 (24.50) | 61.87 (27.34) | 60.43 (25.04)
  Like - Week 4: number analyzed (Participants) | 100 | 110 | 115
  Like - Week 4 | 78.95 (21.61) | 67.78 (25.36) | 69.44 (24.06)
  Enjoy - Week 4: number analyzed (Participants) | 100 | 110 | 115
  Enjoy - Week 4 | 79.16 (20.88) | 68.35 (24.31) | 67.83 (24.41)
  Pleasurable - Week 4: number analyzed (Participants) | 100 | 110 | 114
  Pleasurable - Week 4 | 77.42 (21.82) | 65.95 (24.63) | 67.13 (24.79)
  Satisfying - Week 4: number analyzed (Participants) | 99 | 110 | 114
  Satisfying - Week 4 | 82.17 (17.77) | 63.88 (23.08) | 65.28 (23.28)
  Want - Week 12: number analyzed (Participants) | 98 | 92 | 102
  Want - Week 12 | 71.47 (26.43) | 53.59 (29.50) | 60.45 (26.85)
  Like - Week 12: number analyzed (Participants) | 98 | 93 | 102
  Like - Week 12 | 78.35 (23.58) | 60.71 (30.64) | 67.30 (26.87)
  Enjoy - Week 12: number analyzed (Participants) | 98 | 93 | 102
  Enjoy - Week 12 | 79.49 (21.03) | 60.78 (30.26) | 66.96 (26.59)
  Pleasurable - Week 12: number analyzed (Participants) | 98 | 93 | 102
  Pleasurable - Week 12 | 76.61 (24.13) | 60.27 (30.23) | 65.33 (27.96)
  Satisfying - Week 12: number analyzed (Participants) | 98 | 91 | 102
  Satisfying - Week 12 | 82.12 (19.83) | 57.13 (29.77) | 62.91 (27.94)
  Want - Week 26: number analyzed (Participants) | 55 | 30 | 39
  Want - Week 26 | 72.69 (26.08) | 60.53 (20.04) | 50.23 (22.95)
  Like - Week 26: number analyzed (Participants) | 55 | 30 | 39
  Like - Week 26 | 75.96 (25.42) | 66.53 (23.86) | 67.33 (24.79)
  Enjoy - Week 26: number analyzed (Participants) | 55 | 30 | 39
  Enjoy - Week 26 | 71.91 (27.88) | 68.27 (18.79) | 65.36 (25.56)
  Pleasurable - Week 26: number analyzed (Participants) | 55 | 30 | 39
  Pleasurable - Week 26 | 76.58 (22.94) | 70.20 (19.39) | 61.59 (24.79)
  Satisfying - Week 26: number analyzed (Participants) | 55 | 30 | 39
  Satisfying - Week 26 | 79.73 (20.66) | 68.73 (20.65) | 60.79 (24.73)
  Want - Week 52: number analyzed (Participants) | 50 | 11 | 13
  Want - Week 52 | 67.56 (23.57) | 64.55 (24.79) | 49.23 (29.38)
  Like - Week 52: number analyzed (Participants) | 50 | 11 | 13
  Like - Week 52 | 71.52 (24.39) | 74.09 (24.09) | 67.46 (17.28)
  Enjoy - Week 52: number analyzed (Participants) | 50 | 11 | 13
  Enjoy - Week 52 | 74.36 (21.95) | 73.18 (27.13) | 65.54 (20.41)
  Pleasurable - Week 52: number analyzed (Participants) | 50 | 11 | 13
  Pleasurable - Week 52 | 72.12 (22.78) | 71.00 (26.65) | 61.08 (19.38)
  Satisfying - Week 52: number analyzed (Participants) | 50 | 11 | 13
  Satisfying - Week 52 | 77.96 (21.63) | 74.82 (25.42) | 65.00 (17.70)

7. Secondary Outcome: Biomarker of Exposure - NNAL
Description: Urinary total 4-(methylnitrosamine)-1-(3-pyridyl)-1-butanol [NNAL] (ng/g creatinine)
Time Frame: Baseline, Week 4, Week 12
Reporting Status: Not Posted, anticipated posting 2025-11

8. Secondary Outcome: Biomarker of Exposure - NNN
Description: Presence of urinary [pyridine-D4]NNN ([D4]NNN)
Time Frame: Baseline, Week 4, Week 12
Reporting Status: Not Posted, anticipated posting 2025-11

9. Secondary Outcome: Biomarker of Exposure - Total Nicotine Equivalents (TNE)
Description: Sum of nicotine and metabolites in urine
Time Frame: Baseline, Week 4, Week 12
Reporting Status: Not Posted, anticipated posting 2025-11

10. Secondary Outcome: Biomarker of Exposure - Nicotine Metabolite Ratio
Description: Biomarker of nicotine clearance formed using the ratio of 2 nicotine metabolites (3'hydroxycotinine [3HC]/cotinine)
Time Frame: Baseline, Week 4, Week 12
Reporting Status: Not Posted, anticipated posting 2025-11

11. Secondary Outcome: Biomarker of Exposure - Nickel and Other Relevant Metals
Description: Metals and metalloids in saliva
Time Frame: Baseline, Week 4, Week 12
Reporting Status: Not Posted, anticipated posting 2025-11

12. Secondary Outcome: Biomarker of Exposure - Cadmium and Other Relevant Metals
Description: Metals and metalloids in saliva
Time Frame: Baseline, Week 4, Week 12
Reporting Status: Not Posted, anticipated posting 2025-11

13. Secondary Outcome: Biomarker of Exposure - Lead and Other Relevant Metals
Description: Metals and metalloids in saliva
Time Frame: Baseline, Week 4, Week 12
Reporting Status: Not Posted, anticipated posting 2025-11

14. Secondary Outcome: Biomarker of Exposure - 8-iso-PGF2a
Description: Urinary biomarker of oxidative stress and inflammation
Time Frame: Baseline, Week 4, Week 12
Reporting Status: Not Posted, anticipated posting 2025-11

15. Secondary Outcome: Biomarker of Exposure - PGEM
Description: Urinary biomarker of oxidative stress and inflammation
Time Frame: Baseline, Week 4, Week 12
Reporting Status: Not Posted, anticipated posting 2025-11

16. Secondary Outcome: Biomarker of Effect - q-PADDA
Description: Data is shown as change in DNA damage from baseline. We calculated change in DNA damage in Transcribed (TS) and Non-transcribed strand (NTS) and added those data points to calculate the Total Change in DNA damage.
Time Frame: Week 4, Week 12
Reporting Status: Not Posted, anticipated posting 2025-11

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Usual Brand Cigarette | Low Wattage E Cigarette Device | High Wattage E Cigarette Device
All-Cause Mortality (participants affected / at risk) | 0/105 | 0/133 | 0/134
Serious Adverse Events (participants affected / at risk) | 3/105 | 2/133 | 2/134
Other Adverse Events (participants affected / at risk) | 64/105 | 103/133 | 95/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Brand Cigarette (N=105) | Low Wattage E Cigarette Device (N=133) | High Wattage E Cigarette Device (N=134)
Stroke (Cardiac disorders) | 1 | 0 | 0
High Blood Pressure (Cardiac disorders) | 1 | 0 | 0
Blood Clot (Cardiac disorders) | 1 | 0 | 0
Possible Skin Cancer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Heart Attack (Cardiac disorders) | 1 | 0 | 0
Heartburn (Gastrointestinal disorders) | 0 | 1 | 0
Knee Surgery (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0
Loss of feeling in mouth and jaw (Nervous system disorders) | 0 | 0 | 1
Sharp Chest Pains (Cardiac disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Brand Cigarette (N=105) | Low Wattage E Cigarette Device (N=133) | High Wattage E Cigarette Device (N=134)
Allergies (Immune system disorders) | 9 | 13 | 10
Breathing Difficulties (Respiratory, thoracic and mediastinal disorders) | 23 | 24 | 23
Chest Pain (General disorders) | 3 | 7 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 58 | 68 | 78
Dizziness (Nervous system disorders) | 9 | 14 | 13
Sore or Dry Mouth and Throat (Gastrointestinal disorders) | 25 | 44 | 46
Gingivitis (Gastrointestinal disorders) | 5 | 11 | 7
Headache (Nervous system disorders) | 10 | 18 | 23
Mouth or Tongue Sores / Inflammation (Gastrointestinal disorders) | 2 | 7 | 10
Sleepiness (Nervous system disorders) | 7 | 7 | 9
Sleeplessness (Psychiatric disorders) | 15 | 12 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-20): https://cdn.clinicaltrials.gov/large-docs/36/NCT03113136/Prot_SAP_000.pdf